CLINICAL TRIAL: NCT03376438
Title: FAST Trial Registry: Prospective Observational Cohort Study of Fetal Atrial Flutter & Supraventricular Tachycardia
Brief Title: Prospective Observational Cohort Study of Fetal Atrial Flutter & Supraventricular Tachycardia
Acronym: FAST Registry
Status: Completed | Type: Observational
Sponsor: Edgar Jaeggi (Other)
Responsible Party: Sponsor-Investigator, Edgar Jaeggi, Senior Associate Scientist Emeritus Edgar Jaeggi, MD FRCPC, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Other Study IDs: 1000048953
Record Dates: First submitted 2017-09-27; First posted 2017-12-18 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-04

CONDITIONS: Atrial Flutter; Tachycardia, Supraventricular; Tachycardia, Atrial Ectopic; Tachycardia, Reciprocating; Tachycardia Atrial; Tachycardia, Atrioventricular Nodal Reentry; Tachycardia, Paroxysmal; Fetal Hydrops
MeSH Terms: conditions — Atrial Flutter; Tachycardia, Supraventricular; Tachycardia, Ectopic Atrial; Tachycardia, Reciprocating; Tachycardia, Atrioventricular Nodal Reentry; Tachycardia, Paroxysmal; Hydrops Fetalis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prospective observational cohorts: 1) Atrial flutter without fetal hydrops; 2) Atrial flutter with fetal hydrops; 3) Supraventricular tachycardia without fetal hydrops; and 4) Supraventricular tachycardia with fetal hydrops
  Interventions: Other: Prospective observational cohorts

INTERVENTIONS:
Other: Prospective observational cohorts — Patients with AF or SVT that is significant enough to consider prenatal treatment are eligible for enrollment. Management decisions are made at each patient encounter by the primary physician based on clinical findings and may include: 1) no antiarrhythmic treatment; 2) transplacental antiarrhythmic treatment; 3) direct fetal antiarrhythmic treatment; 4) delivery. Patients enrolled in the FAST Registry will be followed from the time of enrollment until the baby is discharged after birth.
  Other Names: Non-randomized antiarrhythmic fetal drug therapy

SUMMARY:
The FAST Trial Registry is a prospective observational cohort study of fetuses with a new diagnosis of atrial flutter (AF) or supraventricular tachycardia (SVT) that is severe enough to consider prenatal treatment (see eligibility criteria below). Aims of the Registry include to establish a large clinical database to determine and compare the efficacy and safety of different prenatal treatment strategies including observation without immediate treatment, transplacental antiarrhythmic fetal treatment and direct fetal treatment from the time of tachycardia diagnosis to death, neonatal hospital discharge or to a maximum of 30 days after birth.

DETAILED DESCRIPTION:
Few studies are specifically designed to address health concerns relevant during pregnancy. The consequence is a lack of evidence on best clinical practice. This includes mothers and their babies when pregnancy is complicated by an abnormally fast heart rate up to 300 beats per minute due to supraventricular tachyarrhythmia (SVA) in the unborn baby (fetus). Although fetal SVA, including AF and other forms of SVT, is the most common cause of intended in-utero fetal therapy, our knowledge of drug effects on the baby and the co-treated mother is still limited. The Fetal Atrial Flutter and Supraventricular Tachycardia (FAST) Therapy Trial is a prospective multi-center trial to address this knowledge gap in order to guide future patient management to the best of care.

FAST Trial components include:

1. A prospective Registry (FAST Registry; see this document) as well as
2. Three prospective Randomized Clinical Trials (FAST RCTs; see ClinicalTrials.gov #NCT02624765).

The FAST Registry is a prospective observational cohort study to determine the impact of different prenatal treatment strategies on patients diagnosed with fetal AF without hydrops, AF with hydrops, SVT without hydrops, and SVT with hydrops. All management decisions including the choice of antiarrhythmic medication or the decision to observe without treatment are at the discretion of the treating physician. The primary outcome measure will be the proportion of term deliveries of live-born children with a normal cardiac rhythm. Secondary outcome measures include the efficacy of 1st line, 2nd line, 3rd line, and maintenance drug therapy in controlling the different arrhythmias prior to birth and patient safety.

Participation of a site in the FAST Registry requires experience with the perinatal management of fetal AF and SVT, local REB/IRB approval and an executed legal contract with the Hospital for Sick Children, Toronto.

Participation of a patient in the FAST Registry requires that all inclusion and none of the exclusion criteria are fulfilled (see below). Enrollment is possible within 2 days of the arrhythmia diagnosis and the initial management decision.

ELIGIBILITY:
Inclusion Criteria:

1. Mother has provided written informed consent to participate
2. Fetal AF or SVT with or without hydrops
3. Tachyarrhythmia that is significant enough to justify immediate transplacental pharmacological treatment:

   * Tachycardia ≥ 180 bpm during at least 10% of observation time of 30 minutes or longer
   * Tachycardia ≥ 170 bpm during +100% of time (≤ 30 0/7 weeks of gestation)
   * Tachycardia ≥ 280 bpm (irrespective of SVA duration)
   * SVT with fetal hydrops (irrespective of duration)
4. Gestational age <36 0/7 weeks at time of enrollment
5. Singleton Pregnancy
6. Healthy mother with ± normal pre-treatment cardiovascular findings:

   * ECG within normal range (sinus rhythm; QTc ≤ 0.47; PR ≤ 0.2 sec; QRS: ≤ 0.12 sec; insignificant anomalies; isolated premature beats; isolated complete right bundle
   * Maternal resting heart rate ≥ 50 bpm
   * Maternal systolic BP ≥ 85 mmHg

Exclusion Criteria:

1. Primary delivery for postnatal cardioversion
2. Antiarrhythmic fetal treatment for more than 2 days at time of enrollment
3. Any maternal-fetal conditions associated with high odds of premature delivery and/or death
4. History of significant maternal heart condition (open heart surgery; sick sinus syndrome; long QT, Brugada syndrome; ventricular tachycardia; WPW syndrome; high-degree heart block; cardiomyopathy)

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Enrollment into the Registry is possible within maximally 2 days of the fetal SVA diagnosis and management decision to treat or not to treat. If a mother elects participation in the Registry, her treating physician will continue to provide care in accordance with clinical practice at the site and will decide all therapy including close observation without or with immediate prenatal treatment.
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of live-born children with a delivery at term and a normal cardiac rhythm | Term: 37 0/7 to 41 6/7 weeks

SECONDARY OUTCOMES:
Proportion of patients with cardioversion over time | From date of SVA dignosis until the date of first documented cardioversion or until the date of delivery/fetal death without cardioversion, whichever comes first, assessed up to 30 gestational weeks
  Number of participants with persistent tachycardia compared to number of participants with cardioversion to a normal rhythm over time
Proportion of participants with treatment failure | From date of treatment start until the date of first documented fetal cardioversion or until the date of treatment failure, whichever comes first, assessed up to 30 gestational weeks
  Number of participants with treatment failure compared to number of participants with successful treatment. Treatment failure is defined as one of the following: 1) cross-over to another drug; 2) SVT/AF that persists to birth; 3) preterm birth; 4) death.
Proportion of participants with arrhythmia-related death | From date of arrhythmia diagnosis or date of treatment start to 30 days of life
  Number of participants with arrhythmia-related death compared to other outcomes
Average gestational age at birth | At birth
Birth weight (z-scores; centiles) | At birth
Total days of treatment related maternal and neonatal hospitalizations | From date of diagnosis or treatment begin to 30 days of life
Maternal prevalence of pregnancy/treatment-related AEs and outcomes | Diagnosis to birth
Maternal prevalence of adverse events and outcome | From date of treatment begin to 30 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Jaeggi, MD, FRCPC, Principal Investigator — The Hospital for Sick Children, Toronto, ON, Canada
Locations (41):
- United States (18):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital Colorado, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital, Saint Petersberg, Florida
  - John Ochsner Heart & Vascular Institute, New Orleans, Louisiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Health Care, Minneota, Minnesota
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Cohen Children's Medical Centre/Northwell Health - Lake Success, Lake Success, New York
  - Columbia University, New York, New York
  - Cincinnati Children's Hospital Medical Centre, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Inc Pediatric Cardiology of Austin Practice, Austin, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - West Virginia University Research Corporation, Morgantown, West Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- The Royal Women's Hospital, Melbourne, Australia
- Associação Beneficente Síria - Hospital do Coração, São Paulo, Brazil
- Canada (7):
  - University of Alberta, Edmonton, Alberta
  - The U of British Columbia, Vancouver, British Columbia
  - Alberta Children's Hospital, Calgary, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - CHU Saine-Justine, Montreal, Quebec
- University Hospital Brno, Brno, Czechia
- Pediatric Research Center, Helsinki, Finland
- Centre Hospitalier Universitaire, Grenoble, Alpes, France
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong
- Leiden University Medical Centre, Leiden, Netherlands
- National Medical Research Center for Obstetrics, Gynecology and Perinatology, Moscow, Russia
- Spain (2):
  - BCNatal - Hospital Sant Joan de Deu, Barcelona
  - Hospital Virgen de las Nieves, Granada
- Sweden (3):
  - Queen Silvia Children's Hospital, Göteborg, Skåne County
  - Lund University, Lund
  - Karolinska University Hospital, Astrid Lindgen Childrens Hospital, Solna
- Inselspital Universitatsspital Bern, Bern, Switzerland
- United Kingdom (2):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - St George's University Hospital Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No